CLINICAL TRIAL: NCT06931444
Title: School Based Cohort Study for Myopia-The Beijing Childhood Eye Study
Brief Title: The Beijing Childhood Eye Study
Acronym: BCES
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Beijing Childhood Eye Study; Z201100005520045 (Other Grant/Funding Number: the Science & Technology Project of Beijing Municipal Science & Technology Commission)
Record Dates: First submitted 2025-04-15; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Myopia
Keywords: myopia; child; axial length; refractive error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- grades 1-3 students: Currently enrolled students in grades 1-3 of the selected primary schools, in good health, with normal ocular appearance. All enrolled students have no ocular diseases, no strabismus, ocular trauma, or history of intraocular surgery, with unaided visual acuity of 20/20 or better. Parents consent to participate in the survey and sign informed consent form.

SUMMARY:
Axial myopia has emerged as the leading cause of irreversible vision loss in East Asia, driven by its progression to sight-threatening complications including myopic macular degeneration, retinal detachment, open-angle glaucoma, and other complications. In the current study, we aim to observe the natural course of the development , progression, and its associated factors in children

DETAILED DESCRIPTION:
This is a prospective epidemiological cohort study, recruiting students in grades 1-3 in primary school for myopia. Through stratified cluster random sampling, among aii the primary schools in Dongcheng District, Beijing, schools were stratified into key and ordinary schools, with 2 schools randomly selected from each stratum.

A prospective study cohort comprising 3,667 subjects was established. All study subjects completed a standard questionnaire and underwent routine ophthalmic examinations. Follow-up assessments will be conducted regularly to monitor changes in refractive errors and fundus indicators. Informed consent, approved by the Ethics Committee of Beijing Tongren Hospital, was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria: 1) Currently enrolled students in grades 1-3 of the selected primary schools, in good health, with normal ocular appearance. 2) No ocular diseases, no strabismus, ocular trauma, or history of intraocular surgery, with unaided visual acuity of 20/20 or better. 3) Parental and student consent to participate in the survey and signed informed consent form.

Exclusion Criteria: 1) Not currently enrolled in grades 1-3 of a primary school. 2) Students with pre-existing strabismus, other ocular diseases, or a history of ocular surgery at baseline, or those allergic to cycloplegic eyedrops. 3) Students unable to continue studying at their current school for more than three years from the baseline, including those who transfer to another school or withdraw from the study; 4) parental or student disagreement with participation in the survey.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Grades 1-3 primary school students.
Sampling Method: Non-Probability Sample
Enrollment: 3760 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Myopia development | 3 years
  Myopia was classified as a Spherical equivalent (SE) of -0.5 D or lower, and was further categorized into mild (-3 D < SE ≤ -0.5 D), moderate (-6 D < SE ≤ -3 D), and severe (SE ≤ -6 D). Hyperopia was classified as a SE of +1.0 D or greater. Intermediate refractive states (-0.5 D < SE < +1 D) were considered emmetropic. Astigmatism was defined as an absolute cylinder power of 0.75 diopters (D). Anisometropia were defined by an interocular SE difference of at least 1.0 D.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided